CLINICAL TRIAL: NCT04017637
Title: Resistance Training Intervention to Promote Lean Mass in Youth With IBD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study cancelled
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Margaux J Barnes, PhD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BarnesFDGP2019
Record Dates: First submitted 2019-07-08; First posted 2019-07-12 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Resistance Training; Lean Body Mass; Pediatric
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Parallel 2-arm randomized-controlled pilot trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (UC) (No Intervention): Those randomized to the UC group will complete baseline and post-intervention assessments only. No intervention will be administered.
- Resistance Training Intervention (RT) (Experimental): Those randomized to the RT group will complete baseline and post-intervention assessments at weeks 0 and 12. For the intervention, they will complete resistance training for approximately 12 minutes 2x per week for 12 weeks.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — Static resistance training including two arm and two leg movements will be performed twice per week for 12 weeks.
  Arms: Resistance Training Intervention (RT)

SUMMARY:
Evaluate feasibility, safety, and preliminary estimates of resistance training (RT) efficacy to promote lean body mass accrual in patients with CD aged 14-18. This will be achieved by conducting a parallel 2-arm randomized-controlled pilot trial of RT compared to usual care. At weeks 0 (pre-treatment), 6 (mid-treatment), and 12 (post- treatment), feedback regarding safety, feasibility, and acceptability will be collected from participants through surveys and interviews. Magnitude of the effect size of the intervention on LBM, muscle strength, and health-related quality of life (HRQoL) will also be estimated.

DETAILED DESCRIPTION:
Lean body mass (LBM) deficits are common in Crohn's Disease (CD) and persist beyond achievement of remission. In a recent review of 21 studies with a total of 1,479 youth with Inflammatory Bowel Disease (IBD), 93.6% of patients with CD showed deficits in LBM compared to healthy controls. LBM deficits in CD are multifactorial though largely explained by malnutrition. Even with weight restoration and remission however, youth with CD continue to show deficits in LBM compared to healthy peers. Despite proportional deficits in fat and LBM at baseline, weight restoration is explained by gains in fat without similar gains in LBM, suggesting that additional mechanisms interact to maintain deficits such as low physical activity (PA) or altered energy partitioning. Chronic LBM deficits can have deleterious effects including decreased physical function, myopenia, metabolic dysregulation, increased risk of infection, compromised peak bone mass accrual, and development of osteopenia/osteoporosis. While some factors are not readily modifiable (e.g. underlying disease mechanisms), targeting factors amenable to change may result in an increase in LBM and thus improved health outcomes. Health behaviors, including exercise, are modifiable and associated with the development of LBM. Resistance training (RT) has been associated with improved LBM in youth with and without chronic illness. To our knowledge, no evidence-based resistance training interventions have been developed to promote LBM accrual in pediatric CD. The overarching aims of this proposal are to evaluate the safety, feasibility, and effects of 12 weeks of RT on LBM in youth with CD aged 14-18. Specifically we aim to:

Aim 1: Evaluate feasibility, safety, and preliminary estimates of RT efficacy to promote LBM accrual in patients with CD aged 14-18. This will be achieved by conducting a parallel 2-arm randomized-controlled pilot trial of RT compared to usual care. At weeks 0 (pre-treatment), 6 (mid-treatment), and 12 (post- treatment), feedback regarding safety, feasibility, and acceptability will be collected from participants through surveys and interviews. Magnitude of the effect size of the intervention on LBM, muscle strength, and health-related quality of life (HRQoL) will also be estimated.

Positive findings would have broad implications for growth and long-term health outcomes including bone disease and metabolic health in these young patients. More broadly, the findings would have promising potential to be extended to patients with IBD across the developmental and disease spectrum including youth with ulcerative colitis (UC) and adults with IBD as they demonstrate similar LBM deficits. The proposed study will also provide preliminary data to inform a evaluation through a larger trial.

ELIGIBILITY:
Inclusion Criteria.

* aged 14-18
* diagnosed with Crohn's Disease
* able to read, write, and speak English
* have a consenting caregiver who can commit to all study procedures
* have clearance from their primary treating IBD physician to enroll in the RT intervention

Exclusion Criteria:

* history of neuro-developmental or neuro-motor disorder (including but not limited to Intellectual Disability, Down Syndrome, or Cerebral Palsy)
* presence of another medical condition that prevents them from being able to participate in physical activity
* currently participating in a formal exercise or physical activity program beyond physical education offered at school
* currently on systemic steroids

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Change in body composition as measured by DEXA | 12 weeks
Change in muscle strength as measured using a hand dynamometer | 12 weeks
Change in Health-related quality of life as measured by the PedsQL4.0 | 12 weeks

SECONDARY OUTCOMES:
Change in Disease Activity as measured by C-reactive protein blood test | 12 weeks

OTHER OUTCOMES:
Total number of intervention sessions attended | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No